CLINICAL TRIAL: NCT01830829
Title: A Multi-center Randomized Placebo Controlled Trial Evaluating the Efficacy of JALYN in Improving Symptoms in Men Diagnosed With Benign Prostatic Hyperplasia (BPH) and Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Brief Title: JALYN for Benign Prostatic Hyperplasia (BPH) and Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in enrolling particpants
Sponsor: Dr. J. Curtis Nickel (Other)
Collaborators: The Cleveland Clinic (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Dr. J. Curtis Nickel, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JALYN
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Benign Prostatic Hyperplasia; Chronic Prostatitis
Keywords: BPH; CPPS
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jaylyn (Experimental): Jalyn: dutasteride 0.5 mg/day and tamsulosin 0.4 mg/day combination tablet
  Interventions: Drug: Jalyn
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jalyn — study drug
  Other Names: dutasteride 0.5 mg/day; tamsulosin 0.4 mg/day combination tablet
  Arms: Jaylyn
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Benign Prostatic Hyperplasia (BPH) describes a common medical condition in men over 45 associated with voiding (obstructive) and storage (irritative) lower urinary tract symptoms and is in part related to prostate enlargement and obstruction. The standard medical therapy for this condition includes 5-alpha reductase inhibitors -5ARI (eg dutasteride) or alpha blocker therapy (eg tamsulosin), while the most effective medical therapy for BPH is the combination of these two medications. Approximately 10 to 20% of patients diagnosed with BPH also have either a diagnosis of or symptoms of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) with typical genito-urinary pain and discomfort. This particular subset of patients of BPH patients with prostatitis symptoms pose a therapeutic dilemma. CP/CPPS (organ specific phenotype) is the third most prevalent prostate disease after prostate cancer and BPH. CP/CPPS is very prevalent (3-9% of men) and represents a significant percentage of urology outpatients (3-8% of male outpatient visits)resulting in a major impact on quality of life of patients and economic costs to society. Clinical phenotyping allows for prediction of the patients with CP/CPPS most likely to respond to dutasteride and tamsulosin (age, Lower Urinary Tract Symptoms [LUTS] and prostate related phenotypes [BPH]). It can be estimated that up to 30% of men currently diagnosed with CP/CPPS will include men with co-existing Benign Prostatic Hyperplasia (BPH) We propose to determine the efficacy of JALYN (dutasteride-tamsulosin combination) in the amelioration of prostatitis symptoms in men diagnosed with CP/CPPS who have the following clinical phenotype; age = 45 years, Lower Urinary Tract Symptoms (LUTS), enlarged prostate and Organ (prostate) specific symptoms (eg. BPH and CP/CPPS).

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) describes a common medical condition in men over 45 associated with voiding (obstructive) and storage (irritative) lower urinary tract symptoms and is in part related to prostate enlargement and obstruction [1]. The standard medical therapy for this condition includes 5-alpha reductase inhibitors -5ARI (eg dutasteride) or alpha blocker therapy (eg tamsulosin), while the most effective medical therapy for BPH is the combination of these two medications [2]. Approximately 10 to 20% of patients diagnosed with BPH also have either a diagnosis of or symptoms of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) with typical genito-urinary pain and discomfort [3,4,5]. This particular subset of patients of BPH patients with prostatitis symptoms pose a therapeutic dilemma [6].

CP/CPPS (organ specific phenotype) is the third most prevalent prostate disease after prostate cancer and BPH. CP/CPPS is very prevalent (3-9% of men) [7,8] and represents a significant percentage of urology outpatients (3-8% of male outpatient visits) [9,10] resulting in a major impact on quality of life of patients [11] and economic costs to society [12].

There are no good evidence based therapies for CP/CPPS [13,14], although there is some evidence available to consider 5 alpha reductase inhibitor and alpha blocker therapies [22]. There is an enormous unmet need to evaluate potential therapies for this condition.

Our current understanding of CP/CPPS patients are that they are a heterogeneous group of unique patients (the "snow flake" hypothesis) presenting with different clinical phenotypes [15]. We have proposed [16,17], validated [18] and recently proved that clinical phenotyping (using our UPOINT classification system) is possible and provides more effective treatment strategies [19].

There are studies that suggest that the same medical therapy that has proven effective for the treatment of BPH would also be beneficial for prostatitis like symptoms as well. A number of small pilot studies with finasteride [20], including a contemporary 6 month RCT [21], have strongly suggested that 5 ARI therapy may be effective in patients with CP/CPPS, but these studies were limited by study design including inclusion of all patients with the diagnosis of CP/CPPS (ages and clinical phenotypes that we now know could not possibly benefit from a 5ARI). REDUCE and many other epidemiology studies, have documented that men over 45 years old suffer from prostatitis and prostatitis symptoms [23]. REDUCE also clearly shows that dutasteride favorably impacts on prostatitis-like symptoms and men with prostatitis-like syndrome enrolled in that study [24]. In fact, the potential benefits suggested by extrapolating REDUCE results far outweigh any other intervention we have evaluated in any of the large North American NIH sponsored RCTs in the last decade [25,26,27]. A further sub-analyses of REDUCE shows that men with IPSS ≥ 8 and enlarged prostates (eg BPH) have a significant symptom benefit with dutasteride, irregardless of prostate size [28].These initial findings in REDUCE in patients not specifically diagnosed with CP/CPPS should be expanded to examine the benefits in a CP/CPPS population.

There are more clinical trials evaluating alpha blockers than any other therapy in CP/CPPS [22, 29]. While two North American RCTs [25,26] did not show benefit, 6 other alpha blocker randomized placebo controlled trials using validated contemporary outcomes were positive in terms of measureable benefits [30-35]. The latest clinical trial confirming the benefits of alpha blocker therapy in selected CP/CPPS patients (approximately 50 patients per arm in 12 week study) was recently published [35] and showed benefit, primarily in the LUTS symptom domain.

Clinical phenotyping allows for prediction of the patients with CP/CPPS most likely to respond to dutasteride and tamsulosin (age, Lower Urinary Tract Symptoms [LUTS] and prostate related phenotypes [BPH]). It can be estimated that up to 30% of men currently diagnosed with CP/CPPS will include men with co-existing Benign Prostatic Hyperplasia (BPH)

ELIGIBILITY:
Inclusion Criteria:

Men will be eligible for the study if:

1. age at least 45 years
2. report symptoms of discomfort or pain in the pelvic region during at least 3 of the previous 6 months
3. total score of at least 12 (out of 43) points on the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) at both a screening and randomization visit
4. IPSS score of at least 8 points 5 tenderness on light palpation of the prostate

6. prostate size estimated to be at least 30cc on digital rectal examination

Exclusion Criteria:

Participants are excluded if

1. prior treatment with dutasteride or finasteride. Alpha blocker therapy within 3 months of randomization.
2. documented urinary tract infection (>105 colony forming units per ml of a recognized uropathogen)
3. history of renal failure (or calculated creatinine clearance of < 60 ml/min)
4. symptomatic genital herpes in the last 3 months.
5. unilateral orchalgia without pelvic symptoms
6. a history of active urogenital cancer
7. active urethral stricture.
8. surgery of the lower urinary tract (not including simple diagnostic cystoscopy) in the previous 6 months (including TURP, bladder neck incision, bladder tumor resection, urethrotomy).
9. History of alcohol abuse
10. neurologic disease affecting voiding or the bladder
11. Psychiatric condition that would make it difficult (in opinion of investigator) for patient to participate in the study
12. Other acute or chronic medical condition that would make it difficult (in opinion of investigator) for patient to participate in the study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Chronic Prostatitis Symptom Index (CPSI) | 6 months
  The primary endpoint will be the mean change in NIH CPSI from baseline in the treated group compared to the mean change in NIH CPSI from baseline in the placebo group at 6 months.

SECONDARY OUTCOMES:
Pain subdomain | 6 months
  Secondary endpoints will include analyses of CPSI subdomains (pain, urinary, quality of life)
IPSS | 6 months
  International Prostate Symptom Score changes (IPSS)from placebo
GRA | 6 months
  Seven point Global Response Assessment (GRA) where responders will be defined as those who report a moderate or marked improvement.
Urinary subdomain | 6 months
  Secondary endpoints will include analyses of CPSI subdomains (pain, urinary, quality of life)
Quality of Life subdomain | 6 months
  Secondary endpoints will include analyses of CPSI subdomains (pain, urinary, quality of life)

OTHER OUTCOMES:
Safety | 6 months
  Examination of AE and SAEs numbers

CONTACTS AND LOCATIONS:
Overall Officials: J. Curtis Nickel, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Applied Urological Research, Kingston, Ontario, Canada